CLINICAL TRIAL: NCT07009158
Title: Ketamine Assisted Psychotherapy to Improve Quality of Life in Veterans and Civilians With Comorbid Chronic Pain and Posttraumatic Stress Disorder: an Open-label Randomized Controlled Trial.
Brief Title: Ketamine Assisted Psychotherapy for Treating Comorbid Chronic Pain and PTSD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Kingston Health Sciences Centre (Other); Providence Care Hospital, Kingston, ON, Canada (Unknown)
Responsible Party: Principal Investigator, Tim Salomons, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAQ-6043701
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Posttraumatic Stress Disorder (PTSD)
Keywords: Ketamine; Mindfulness-based Cognitive Therapy
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KAP group (Experimental): The Ketamine-assisted psychotherapy (KAP) group will receive 4 ketamine infusion treatments and 8 sessions of mindfulness therapy.
  Interventions: Drug: Ketamine Infusion; Behavioral: Mindfulness-based cognitive therapy
- MT group (Active Comparator): The mindfulness therapy (MT) group will receive only the psychotherapy treatment (8 sessions mindfulness therapy).
  Interventions: Behavioral: Mindfulness-based cognitive therapy

INTERVENTIONS:
Drug: Ketamine Infusion — Ketamine hydrochloride (DIN: 02246795, 02246796) will be administered over 40-min intravenous (IV) infusion twice per week on non-consecutive days for the first two weeks of study treatment (four treatment sessions in total). We will use a standard dose of 0.5mg/kg which has demonstrated efficacy in safety in individuals with PTSD.
  Arms: KAP group
Behavioral: Mindfulness-based cognitive therapy — The Mindfulness-based cognitive therapy (MBCT) will be an 8-week group program adapted from a protocol developed to treat PTSD to include psychoeducation about chronic pain and mutual maintenance factors through which chronic pain and PTSD facilitate each other. The MBCT group will be delivered by trained professionals in weekly 2-hour sessions through Microsoft Teams. The 8-week program will include 1) mindfulness techniques; 2) psychoeducation regarding chronic pain, PTSD and stress responses; 3) psychoeducation on mutual maintenance factors that contribute to negative interactions between pain and PTSD symptoms, 4) promoting mindful awareness of these factors' impact on daily life and 5) feedback and supportive group discussion of exercises. Participants will be asked to complete daily mindfulness exercises between sessions to practice skills learned for a recommended minimum of 20 minutes per day.

SUMMARY:
The goal of this pilot study is to evaluate the feasibility of conducting a clinical trial assessing if ketamine infusions combined to mindfulness therapy works better than psychotherapy alone to treat chronic pain and PTSD in adults living with both conditions. The objectives of the pilot study are to 1) assess the feasibility of the trial methods and 2) assess the feasibility and tolerability of ketamine treatment in combination with psychotherapy. The main questions the future full trial would aim to answer are:

* Does the combination of ketamine infusion treatment and mindfulness therapy improve the quality of life in adults living with both chronic pain and PTSD more effectively than mindfulness therapy alone?"
* Does the combination of ketamine infusion treatment and mindfulness therapy improve disability, and depressive, PTSD and pain symptoms in adults living with both chronic pain and PTSD more effectively than mindfulness therapy alone?"
* Does implementing a brief ketamine infusion protocol safe and tolerable to treat chronic pain and PTSD?

Researchers will compare ketamine infusion treatment combined with mindfulness therapy to mindfulness therapy alone to see if the combined treatment works better to treat chronic pain and PTSD.

Participants will:

* Attend 6 visits with a research team member to complete assessments and questionnaires.
* Attend 4 ketamine treatment over 2 weeks, if allocated to the experimental group.
* Attend 8 mindfulness therapy group sessions online (1 per week).
* Log mindfulness exercises completed during the study period.

ELIGIBILITY:
Inclusion Criteria:

i) A current DSM-5 diagnosis of PTSD (confirmed by the Mini International Neuropsychiatric Interview (66)) ii) Chronic pain (> 4/10 average pain reported for longer than 3 months (per (67)).

iii) 18-65 years of age. iv) Capacity to consent

Exclusion Criteria:

i) Currently receiving or received ketamine or psychotherapy to treat PTSD in previous 8 weeks.

ii) Meeting DSM-5 criteria for substance abuse disorder within the past month or lifetime history of ketamine abuse.

iii) Concomitant unstable major medical or neurological conditions, or laboratory/imaging results as considered by the study treating physician to interfere with trial participation (e.g. poorly controlled blood pressure, BMI >35).

iv) Pregnancy or the intention to become pregnant and breastfeeding during the study as confirmed by self-report. Participants must be willing to use a medically acceptable method of birth control which include abstinence, hormonal (birth control pills, patch, hormone injections or implants), diaphragm with spermicide or cervical cap, IUD, condom used together with spermicide, surgical sterilization (hysterectomy or partner's vasectomy) and post-menopausal more than 2 years.

v) DSM-5 diagnosis of bipolar disorder, psychotic disorder, or a severe personality disorder which may interfere with the trial. Patients with lifelong diagnosis of Bipolar Disorder, Schizophrenia or Schizoaffective disorder will be excluded. Patients with primary Obsessive Compulsive Disorder, Substance Use Disorder (dependence and abuse), Seasonal Affective Disorder, or Generalized Anxiety Disorder at time of assessment will be excluded. Primary severe borderline personality disorder and any other personality disorders that potentially may interfere with treatment administration will also be excluded.

vi) Deemed to be high suicidal risk during the baseline assessment as per treating physician. Chronic persistent suicidality is not an exclusion.

vii) Use of medications that might interfere with ketamine efficacy such as benzodiazepines with a dose equivalent to lorazepam 2mg/day or higher, and anti-convulsant (except for pregabalin and gabapentin).

viii) Deemed not appropriate to engage in group psychotherapy. ix) Inability to communicate in spoken and written English fluently enough to complete the required study assessments or a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete clinical assessments).

x) Cognitive or physical impairment severe enough to interfere with IV ketamine administration and the subject's ability to stay in the same place for a 2-hr monitoring supervision.

xi) Inability to secure a responsible adult to accompany them back home after ketamine sessions.

xii) Inability to take part in virtual care, no valid email address. xiii) Inability to safely secure IV access.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Enrollment, 1 week pre-treatment, mid-treatment (1month), post-treatment (2months) and follow-up (3months)
  Measured using the Short-Form-12 Health Survey (SF-12v2)

SECONDARY OUTCOMES:
Depressive symptoms | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Measured using the Montgomery-Asberg Depression Rating Scale (MADRS)
Suicide risk | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Suicide risk will be measured using the Columbia-Suicide Severity Rating Scale (C-SSRS)
PTSD symptoms | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Measured using the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5).
Pain Severity | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Pain Severity will be measured using the Brief Pain Inventory - Short Form (BPI)
Pain Interference | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Pain Interference will be measured using the Brief Pain Inventory - Short Form (BPI)
Disability | At enrollment, 1 week pre-treatment, mid-treatment (1 month), post-treatment (2 month), follow-up (3 months)
  Measured using the WHO Disability Assessment Schedule (WHODAS 2.0- 12 items)
Adverse events | From enrollment to 1 month after the end of the 8-week treatment period
  Measured using a adverse events form.

OTHER OUTCOMES:
Baseline Characteristics | Enrollment
  To describe the study population, the investigators will capture the following through the survey: age, sex, gender, duration of pain, locations of pain, current work status, military status, education, income, and ethnicity.
Concomitant medication | At enrollment and follow-up (3 months)
  A list of medication currently used will be provided by the participants. Participants will be asked to talk the the research team before making any changes or start new medications during study period.

IPD SHARING:
Plan to Share IPD: Undecided